CLINICAL TRIAL: NCT05232526
Title: The Effectiveness of Mental Imagery in Motor and Cognitive Rehabilitation in Subjects of Early Stage of Dementia
Brief Title: Imagery in Early Stages of Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of West Attica (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Anna Christakou, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93292 - 26/10/2021
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Mental Imagery; Dementia of Alzheimer Type
Keywords: Imagery; Exercise; Dementia
MeSH Terms: conditions — Motor Activity; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental imagery (MI) and exercise program (Experimental): MI will start immediately when the sample is going to start the exercise program. The intervention group will undergo 24 sessions of imagery, starting from the 1st exercise program session. Participants of the intervention group will undergo a 45-minute imagery session sitting in a quiet place after the end of every exercise program session. The content of every imagery session is alike with the content of the exercise program session. That means that every session includes imagery of the same exercises of the exercise program performed earlier by the subject in the Day Center. Sessions are identical for all subjects of the intervention group. The total duration of the physiotherapy exercise program will be 24 sessions, 2 times/week, duration of 45 minutes each session, 3 months (12 weeks).
  Interventions: Other: Mental imagery (MI) and exercise program; Device: Mental Imagery and Exercise program
- Exercise program (Placebo Comparator): The total duration of the physiotherapy exercise program will be 24 sessions, 2 times/week, duration of 45 minutes each session, 3 months (12 weeks).
  Interventions: Other: Mental imagery (MI) and exercise program

INTERVENTIONS:
Other: Mental imagery (MI) and exercise program — Mental imagery and exercise program will be used to improve balance, functional status, cognitive ability, depression and quality of life of the sample
Device: Mental Imagery and Exercise program — Questionnaires and functional tests are going to be used to evaluate balance, functional status, cognitive ability, depression and quality of life of the sample.
  Arms: Mental imagery (MI) and exercise program

SUMMARY:
The purpose of the present study is to investigate the effectiveness of mental imagery (MI) in subjects with early stage of dementia. The hypothesis of the study is that MI will have a beneficial effect in motor, cognitive and emotional state in this clinical population.

DETAILED DESCRIPTION:
Dementia is a disorder that is characterized by a decline in cognition involving one or more cognitive domains (learning and memory, language, executive function, complex attention, perceptual-motor, social cognition). The most common form of dementia in older adults is Alzheimer disease (AD), accounting for 60 to 80 percent of cases.

Mental imagery (MI) is a technique which involves envisioning motor actions without actual execution. MI is considered an effective rehabilitative tool in athletes, Parkinson's disease, and post stroke because it engages the same or similar neural systems as the actual execution of motor actions to improve gait, gait-related, and cognitive functions having as a result improvements in gait speed, stride length, tandem stance, timed up and go, clock drawing and stroop interference.

The recruitment of the population will be carried out by Day Care Centers in Athens Alzheimer Association. A group of elderly patients with early stage of dementia, aged 65 to 95 years, will participate. Information sheet and consent form will be provided to all participants. A randomized intervention study is designed to assess the efficacy of MI as therapeutic strategy for subjects with early stage of dementia and the sample will be randomized to one of the three following study groups: 1. MI and exercise program (intervention group) 2. Only exercise program (control group) 3. Neither MI nor exercise program (2nd control group). Assessment will be obtained in three-time periods: prior to the program, middle of the program and after the program.

ELIGIBILITY:
Inclusion Criteria:

* 95 years<age>65 years
* Diagnosed early stage of dementia
* Good oral and written speech and to perform orders
* Both sexes
* Ambulatory
* No other health issues in the last month

Exclusion Criteria:

* Late stage of dementia
* Psychiatric problems
* Serious health problems
* Not able to walk

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Change is being assessed (Change from Baseline Balance at 12 weeks) | Prior to the 1st week of the program, the 12th week of the program
  The Berg Balance Scale (BBS) is used to objectively determine a subject's ability to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a 5-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Change is being assessed (Change from Baseline Stability at 12 weeks) | Prior to the 1st week of the program, the 12th week of the program
  The Multidirectional Reach Test (Reach in Four Directions Test) is a screening tool to determine the limits of stability of subjects in 4 directions: forward, backward, leftward and rightward. Subjects performed maximal outstretched arm reach in each direction with their feet flat on the floor.
Change is being assessed (Change from Baseline Siti-to-stand ability at 12weeks) | Prior to the 1st week of the program, the 12th week of the program
  The Five Times Sit-to-Stand Test (FTSST) is considered to be a useful, consistent and low-cost tool to assess sit-to-stand ability. The FTSST measures the time taken to stand five times from a sitting position as quickly as possible that measures of lower limb strength, balance control and exercise capacity.
Change is being assessed (Change from Baseline Functional status at 12 weeks) | Prior to the 1st week of the program, the 12th week of the program
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility. It measures the time that a subject takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.

SECONDARY OUTCOMES:
Cognitive ability | Prior to the 1st week of the program, the 6th week of the program, the 12th week of the program
  The Walking While Talking Test (WWITT) is a dual-task measure to examine cognitive-motor interactions. During the WWTT, subjects walk at self-paced speed for 6 meters before turning and walking back to the starting point. During the walking subjects recite 12 Greek alphabet letters (each letter at each step) starting with "A" (ΑΒΓΔ, ΚΛΜΝ, ΠΡΣΤ) until the starting point. Time and errors in the alphabet will be recorded.
Depression | Prior to the 1st week of the program, the 6th week of the program, the 12th week of the program
  The Short-Form of Geriatric Depression Scale (SF-GDS) is a 15-question screening tool for depression in older adults, using a "Yes/No" format. It takes 5-7 minutes to complete and is filled out by the researcher with minimal training in its use.
Quality of life | Prior to the 6th week of the program, the 6th week of the program, the 12th week of the program
  The Euro-Qol 5 Dimensions 5 Level of severity scale (Euro-Qol 5D-5L scale) is a preference-based Health Related Quality of Life measure which includes 5 domains, i.e., mobility, self-care, usual activities, pain/discomfort, anxiety/depression. The core of all domains ranges from 1 (best score) up to 5 (worse score). The total perceived quality of life will be graded by the patient. Also it includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Locations (1):
- University of West Attica, Athens, Aigaleo, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christakou A, Bouzineki C, Pavlou M, Stranjalis G, Sakellari V. The effectiveness of mental imagery on motor, cognitive and emotional status of older people with early-stage dementia: A study protocol. J Frailty Sarcopenia Falls. 2023 Mar 1;8(1):60-65. doi: 10.22540/JFSF-08-060. eCollection 2023 Mar. PMID 36873828